CLINICAL TRIAL: NCT03184935
Title: Research for Human Umbilical Cord Mesenchymal Stem Cells in the Treatment of Myelodysplastic Syndrome (MDS)
Brief Title: Research for Human Umbilical Cord Mesenchymal Stem Cells (19#iSCLife®-MDS) in the Treatment of Myelodysplastic Syndrome (MDS)
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Others
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCLnow-IMIMH-03
Record Dates: First submitted 2017-06-06; First posted 2017-06-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; mesenchymal stem cells
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Basic medication: Decitabine; Allogeneic umbilical cord mesenchymal stem cells.
  Interventions: Biological: Allogeneic umbilical cord mesenchymal stem cells; Drug: Decitabine
- Control group (Placebo Comparator): Basic medication: Decitabine; placebo: saline.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Biological: Allogeneic umbilical cord mesenchymal stem cells — Experimental group receive Allogeneic umbilical cord mesenchymal stem cell，i.v (SCLnow 19#)
  Arms: Experimental group
Drug: Decitabine — Decitabine，20mg/m^2/d

SUMMARY:
The purposes of the study is to determine the safety and efficacy of human umbilical cord mesenchymal stem cells (hUC-MSC) in treating Myelodysplastic Syndrome patients.

DETAILED DESCRIPTION:
This is a randomized, double-blind, paralleled study. 40 patients will be separated into two groups, and receive basic treatment (Decitabine). Patients in experimental group will receive hUC-MSC, while control group receive placebo (normal saline), four weeks as a course of treatment. All of the patients accept examination before treatment, including

* diagnostic projects: bone marrow test, peripheral blood classification, chromosome, and MDS fusion gene test, etc.;
* routine examination: blood, urine, and stool routine test, X-ray film in chest, electrocardiogram, etc.;
* stem cell-based medicinal products usage, dosage, time, and course of treatment.

Then, patients will accept routine examination everyday, and after treatment, investigator will follow-up for 6 months, to evaluate the security and efficacy of hUC-MSC.

ELIGIBILITY:
Inclusion Criteria:

* MDS patients with international prostate symptom score is moderate or severe symptoms

Exclusion Criteria:

* with serious renal function impaired
* with other organ function abnormal: acute hepatitis B, ejection fraction < 40%, serum bilirubin > 3mg/dl, liver function tests abnormal, central nervous system disease, mental disease
* bad physical condition (Karmofsky < 60%)
* without signing informed consent form
* under other therapy that possibly influence MSC security or efficacy
* HIV or other serious disease infection
* Donor: HIV, active hepatitis B/C infection, Syphilitic antibody positive
* Donor/ participants: alcoholism, drug addicted, mental disease

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment related-adverse events counting | 16 weeks
  patients will be monitored for any adverse events resulting from the treatment of Human Umbilical Cord Mesenchymal Stem Cells

SECONDARY OUTCOMES:
Improvement in clinical function | 16 weeks
  According to 'Diagnostic and Curative Criteria of Hematological Diseases' 3rd edition edited by Zhang Zhinan and Shen Di, evaluate the hUC-MSCs efficacy. The result as follow:
  * complete remission (CR);
  * partial remission (PR);
  * stable disease (SD);
  * progressive disease (PD)

CONTACTS AND LOCATIONS:
Overall Officials: Shana Chen, Study Director — Inner Mongolia International Mongolian Hospital; Lei Guo, Study Chair — China-Japan Union Hospital, Jilin University
Locations (1):
- Inner Mongolia International Mongolian Hospital, Hohhot, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: No